CLINICAL TRIAL: NCT06190977
Title: Effects of the Otago Exercise Program on Rehabilitation Outcomes of Balance, Strength and Functional Outcomes in Post-Operative Total Knee Replacement Patients
Brief Title: Effects of OEP on Rehabilitation Outcomes on TKR Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Farrah azeem
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Total Knee Replacement
Keywords: Otago Exercise Program; balance; strength; osteoarthritis; ADLs
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Otago Exercise Program (Experimental): Warm-up activities for 5 min head movement, neck movement, back stretching, trunk movement, and ankle movement.
  strength and balance training for 30 mins Strengthening training include sitting knee extension, standing hip abduction, standing knee flexion, tiptoe and heel tiptoe Balance training include standing on one foot, walking in the shape of the number eight, walking sideways, walking backward, standing to sit position training, knee bending, toe to heel standing, heel walking, toe to heel walking, toe to heel walking, toe to heel walking, toe to heel walking backward, and climbing stairs Walking training for 10 min
  Interventions: Other: Otago Exercise Program
- General TKR ptotocol (Other): Ankle pumps Straight leg raises Heel slides Seated knee extensions Standing knee flexion Calf raises Quadriceps contraction Stationary bike
  Interventions: Other: General TKR pprotocol

INTERVENTIONS:
Other: Otago Exercise Program — Exercises will include Intensity: 10 repetitions of each set for the first two weeks and 15 repetitions of each set for the last two weeks, Frequency 3 sessions per week for 4 weeks. Time= 40-45 minutes
  Arms: Otago Exercise Program
Other: General TKR pprotocol — Exercises will include Intensity: 10 repetitions of each set, Frequency 5 sessions per week for 4 weeks. Time= 30 minutes
  Arms: General TKR ptotocol

SUMMARY:
The aim of this research is to assess the effects of the Otago Exercise Program on Rehabilitation outcomes of balance strength and functional outcomes of post Total Knee Replacement patients. A randomized controlled trial that will include a total of 44 participants divided into two groups control and experimental. The experimental group will receive the Otago Exercise Program for four weeks, three times per week for forty to forty-five minutes. The control group will receive general TKR protocol for four weeks, three times per week for 30 minutes. Data collected will be analyzed through SPSS 25.

DETAILED DESCRIPTION:
Total knee replacement (TKR) is one of the most effective surgical interventions for the relief of pain and functional recovery in patients with advanced osteoarthritis (OA) of the knee. In this procedure, the knee joint is resurfaced with a metal or plastic implant intended to restore function, provide pain relief, and improve quality of life.

According to a study in Pakistan, a total of 14,875 people had total knee replacement in the last seven years from 2014 to 2021 with a rate of 14.8/100,000 population. In the United States, estimates of TKR incidence lie at 400,000 each year, a figure expected to grow 143% by 2050 even through conservative projections.

TKR is considered one of the most effective procedures in orthopedic surgery, but electing for it is far from straightforward: noninvasive alternatives such as weight loss, physical therapy, and NSAIDs are first exhausted. If unsuccessful, a patient will undergo a thorough examination of clinical history and comprehensive imaging of the joint to determine if a TKR is feasible, and if so, the desired implant design and size.

Despite the improvements in surgical techniques, the outcomes after TKR remain strongly influenced by the adequacy of rehabilitation and the consequent functional recovery.

Rehabilitation, with a particular emphasis on physiotherapy and exercise, is widely promoted after TKR. During the hospital stay, physiotherapy targets mobilization and achievement of functional goals relating to hospital discharge. Further post-discharge physiotherapy and exercise-based interventions promote strength and balance re-training and functional improvement. However, the provision of these services varies in content and duration.

However, it has been reported that patients with TKR do not fully recover balance and proprioception in the long-term, remaining clearly below the "abilities" of their healthy matched controls. Low balance and proprioception have been ascribed to the loss of knee receptors located in the structures such as the menisci, the cruciate ligaments, and the cartilage, which are removed for the prosthesis implant.

The Otago Exercise Program (OEP) is a home-based balance and strength training program that reduces falls and promotes muscle strength and balance in daily life.OEP is a multi-modal training method that integrates warm-up exercises (5 movements), progressive muscle strength training (5 movements), balance training (12 movements), walking sessions, and aerobic exercise. Initially, The most significant effects on fall reduction induced by the Otago program were only seen in patients who are 80 years or older but now it has shown promise in diverse rehabilitation contexts. Considering that muscle strength and balance are critical factors of TKR postoperative rehabilitation, it is plausible that postoperative OEP may provide further benefits.

This study will explore the effects of postoperative OEP on rehabilitation outcomes of balance, strength, and functional outcomes in TKR patients in regard to reducing postoperative fall occurrence and enhancing knee function. It is hypothesized that this program (OEP) would be effective with these individuals in accelerating rehabilitation and lowering the risks of falling. We constructed a 4-week intervention plan based on pre-, post and after 2nd week follow-up intervention measures of Otago exercise, and explored more effective intervention strategies of functional exercise after total knee replacement.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Age 45 or above
* 3-6 weeks since replacement surgery
* Berge balance scale 21-40
* Patients should have received medical clearance from their surgeon or health care provider to engage in an exercise program

Exclusion Criteria:

* History of recent musculoskeletal injury of lower limb
* Patients have undergone revision TKR
* Patient with moderate cognitive impairment
* Patients with unstable medical conditions or active infection
* Patient with specific contraindications to exercise as determined by their healthcare provider such as blood clots or severe osteoporosis.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
Berg balance scale | 4th week
  Consists of 14 tasks and total score of 56.score of 0-20 indicates severe fall risk, 20-45 includes moderate risk of fall and 45-60 illustrates thr functional balances state.

SECONDARY OUTCOMES:
timed up and go (TUG) test | 4th week
  The test measures the time it takes for a person to stand up from a chair, walk a short distance (typically 3 meters) turn around, return and sit back down.
short physical performance battery | 4th week
  The test includes three different domains (walking, sit-to-stand and balance) to assess functional mobility. The test is easy to administer and takes approximately 10 mins. The SPPB includes three sub tests.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Aabroo, Nmpt, Principal Investigator — Riphah International University
Locations (1):
- NIRM, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nakano N, Shoman H, Olavarria F, Matsumoto T, Kuroda R, Khanduja V. Why are patients dissatisfied following a total knee replacement? A systematic review. Int Orthop. 2020 Oct;44(10):1971-2007. doi: 10.1007/s00264-020-04607-9. Epub 2020 Jul 8. PMID 32642827
- [Background] Bukhari SI, Allana AR, Najjad KR, Noor SS, Chinoy A. Epidemiology of hip & knee replacement across Pakistan: Multicenter cross-sectional study. Pak J Med Sci. 2023 Nov-Dec;39(6):1557-1561. doi: 10.12669/pjms.39.6.7006. PMID 37936780
- [Background] Tolpadi AA, Lee JJ, Pedoia V, Majumdar S. Deep Learning Predicts Total Knee Replacement from Magnetic Resonance Images. Sci Rep. 2020 Apr 14;10(1):6371. doi: 10.1038/s41598-020-63395-9. PMID 32286452
- [Background] Jester R, Rodney A. The relationship between obesity and primary Total Knee Replacement: A scoping review of the literature. Int J Orthop Trauma Nurs. 2021 Jul;42:100850. doi: 10.1016/j.ijotn.2021.100850. Epub 2021 Feb 16. PMID 34044216
- [Background] Bravi M, Longo UG, Laurito A, Greco A, Marino M, Maselli M, Sterzi S, Santacaterina F. Supervised versus unsupervised rehabilitation following total knee arthroplasty: A systematic review and meta-analysis. Knee. 2023 Jan;40:71-89. doi: 10.1016/j.knee.2022.11.013. Epub 2022 Nov 18. PMID 36410253
- [Background] Hadamus A, Bialoszewski D, Blazkiewicz M, Kowalska AJ, Urbaniak E, Wydra KT, Wiaderna K, Boratynski R, Kobza A, Marczynski W. Assessment of the Effectiveness of Rehabilitation after Total Knee Replacement Surgery Using Sample Entropy and Classical Measures of Body Balance. Entropy (Basel). 2021 Jan 29;23(2):164. doi: 10.3390/e23020164. PMID 33573057
- [Background] de Lima F, Melo G, Fernandes DA, Santos GM, Rosa Neto F. Effects of total knee arthroplasty for primary knee osteoarthritis on postural balance: A systematic review. Gait Posture. 2021 Sep;89:139-160. doi: 10.1016/j.gaitpost.2021.04.042. Epub 2021 Apr 30. PMID 34284334
- [Background] Dominguez-Navarro F, Silvestre-Munoz A, Igual-Camacho C, Diaz-Diaz B, Torrella JV, Rodrigo J, Paya-Rubio A, Roig-Casasus S, Blasco JM. A randomized controlled trial assessing the effects of preoperative strengthening plus balance training on balance and functional outcome up to 1 year following total knee replacement. Knee Surg Sports Traumatol Arthrosc. 2021 Mar;29(3):838-848. doi: 10.1007/s00167-020-06029-x. Epub 2020 Apr 27. PMID 32342139
- [Background] Labanca L, Iovine R, Bragonzoni L, Barone G, Farella GM, Benedetti MG. Instrumented platforms for balance and proprioceptive assessment in patients with total knee replacement: A systematic review and meta-analysis. Gait Posture. 2020 Sep;81:230-240. doi: 10.1016/j.gaitpost.2020.07.080. Epub 2020 Aug 8. PMID 32810699
- [Background] Sun JN, Shan YZ, Wu LX, Li N, Xu FH, Kong XR, Zhang B. Preoperative high-intensity strength training combined with balance training can improve early outcomes after total knee arthroplasty. J Orthop Surg Res. 2023 Sep 15;18(1):692. doi: 10.1186/s13018-023-04197-3. PMID 37715204
- [Background] Chiu HL, Yeh TT, Lo YT, Liang PJ, Lee SC. The effects of the Otago Exercise Programme on actual and perceived balance in older adults: A meta-analysis. PLoS One. 2021 Aug 6;16(8):e0255780. doi: 10.1371/journal.pone.0255780. eCollection 2021. PMID 34358276
- [Background] Peng Y, Yi J, Zhang Y, Sha L, Jin S, Liu Y. The effectiveness of a group-based Otago exercise program on physical function, frailty and health status in older nursing home residents: A systematic review and meta-analysis. Geriatr Nurs. 2023 Jan-Feb;49:30-43. doi: 10.1016/j.gerinurse.2022.10.014. Epub 2022 Nov 19. PMID 36413811
- [Background] Viveiro LAP, Gomes GCV, Bacha JMR, Carvas Junior N, Kallas ME, Reis M, Jacob Filho W, Pompeu JE. Reliability, Validity, and Ability to Identity Fall Status of the Berg Balance Scale, Balance Evaluation Systems Test (BESTest), Mini-BESTest, and Brief-BESTest in Older Adults Who Live in Nursing Homes. J Geriatr Phys Ther. 2019 Oct/Dec;42(4):E45-E54. doi: 10.1519/JPT.0000000000000215. PMID 30407272
- [Background] Demircioglu A, Kezban Sahin U, Acaroz S. Discriminative Ability of the Four Balance Measures for Previous Fall Experience in Turkish Community-Dwelling Older Adults. J Aging Phys Act. 2022 Mar 18;30(6):980-986. doi: 10.1123/japa.2021-0415. Print 2022 Dec 1. PMID 35303710
- [Background] Lauretani F, Ticinesi A, Gionti L, Prati B, Nouvenne A, Tana C, Meschi T, Maggio M. Short-Physical Performance Battery (SPPB) score is associated with falls in older outpatients. Aging Clin Exp Res. 2019 Oct;31(10):1435-1442. doi: 10.1007/s40520-018-1082-y. Epub 2018 Dec 4. PMID 30515724
- [Background] Phu S, Kirk B, Bani Hassan E, Vogrin S, Zanker J, Bernardo S, Duque G. The diagnostic value of the Short Physical Performance Battery for sarcopenia. BMC Geriatr. 2020 Jul 13;20(1):242. doi: 10.1186/s12877-020-01642-4. PMID 32660438